CLINICAL TRIAL: NCT02646878
Title: A Feasibility Study to Evaluate the Performance of the Harmony 1 Sensors in Adults and Pediatrics
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: CEP310
Record Dates: First submitted 2015-12-22; First posted 2016-01-06 (Estimated); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Type 2 Diabetes; Harmony Sensor; Continuous Glucose Monitoring; CGM
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- Harmony 1 Sensor Group A (Other): Subjects wearing Harmony 1 Sensor will be assigned this group which will participate in the in-clinic YSI frequent sample testing 90 minutes after sensor insertion.
  Interventions: Device: Harmony 1 Sensor
- Harmony 1 Sensor Group B (Other): Subjects wearing Harmony 1 Sensor will be assigned this group which will participate in the in-clinic YSI frequent sample testing 12 hours after sensor insertion.
  Interventions: Device: Harmony 1 Sensor

INTERVENTIONS:
Device: Harmony 1 Sensor — Use of Harmony 1 Sensor for 10 days when inserted in the arm and abdomen and used with the Guardian Mobile in subjects aged 14-75 years who have had a diagnosis of type 1 or type 2 diabetes for at least 6 months.

SUMMARY:
The purpose of this study is to demonstrate the performance of the Harmony 1 Sensor in subjects age 14 - 75 years.

DETAILED DESCRIPTION:
The study is a multi-center, prospective single-sample correlational design without controls.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is 14 - 75 years of age at time of screening
2. A clinical diagnosis of type 1 or 2 diabetes for a minimum of 6 months duration as determined via medical record or source documentation by an individual qualified to make a medical diagnosis
3. Adequate venous access as assessed by investigator or appropriate staff

Exclusion Criteria:

1. Subject will not tolerate tape adhesive in the area of Harmony 1 Sensor placement as assessed by qualified individual.
2. Subject has any unresolved adverse skin condition in the area of Harmony 1 Sensor or device placement (e.g., psoriasis, rash, Staphylococcus infection)
3. Subject is actively participating in an investigational study (drug or device) wherein they have received treatment from an investigational study (drug or device) in the last 2 weeks
4. Subject is female and has a positive pregnancy screening test
5. Females of child bearing age and who are sexually active should be excluded if they are not using a form of contraception deemed reliable by investigator
6. Subject is female and plans to become pregnant during the course of the study
7. Subject has had a hypoglycemic seizure within the past 6 months
8. Subject has had hypoglycemia resulting in loss of consciousness within the past 6 months prior to screening visit.
9. Subject has had an episode of diabetic ketoacidosis (DKA) within the past 6 months prior to screening visit.
10. Subject has a history of a seizure disorder
11. Subject has central nervous system or cardiac disorder resulting in syncope
12. Subject has a history of myocardial infarction, unstable angina, coronary artery bypass surgery, coronary artery stenting, transient ischemic attack (TIA), cerebrovascular accident (CVA), angina, congestive heart failure, ventricular rhythm disturbances or thromboembolic disease
13. Subject has a hematocrit (Hct) lower than the normal reference range
14. Subject has a history of adrenal insufficiency.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-01 (Estimated); Primary Completion 2016-07 (Estimated); Study Completion 2016-07 (Estimated)

PRIMARY OUTCOMES:
24 hour calibration requirement | 10 days
  Descriptive summary of sensor accuracy for Harmony 1 Sensor data with the every 24 hour calibration requirements

CONTACTS AND LOCATIONS:
Overall Officials: Ronald Brazg, MD, Principal Investigator — Rainer Clinical Research Center; Mark Christiansen, MD, Principal Investigator — Diablo Clinical Research

IPD SHARING:
Plan to Share IPD: No